CLINICAL TRIAL: NCT01071889
Title: Double-blind, Randomized, Placebo and Active Controlled Study to Assess the Safety and the Efficacy of a Sublingual Administration of Flumazenil to Reverse the Effect of Hypnotic Drugs in Healthy Adults(Zolpidem or Brotizolam)
Brief Title: Safety and the Efficacy of a Sublingual Administration of Flumazenil to Reverse the Effect of Hypnotic Drugs in Healthy Adults
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Coeruleus Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0076-10-RMB
Record Dates: First submitted 2010-02-17; First posted 2010-02-19 (Estimated); Last update posted 2015-01-30 (Estimated); Status verified 2015-01

CONDITIONS: Healthy
Keywords: Healthy Volunteers
MeSH Terms: interventions — Flumazenil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Brotizolam (Other): Treatment response will be evaluated for each treatment arm. Good Response (GR) - is considered as an improvement of 30% in efficacy parameters of Flumazenil treatment in comparison to placebo
  Interventions: Drug: Flumazenil; Drug: Placebo
- Zolpidem (Other): Treatment response will be evaluated for each treatment arm. Good Response (GR) - is considered as an improvement of 30% in efficacy parameters of Flumazenil treatment in comparison to placebo.
  Interventions: Drug: Flumazenil; Drug: Placebo

INTERVENTIONS:
Drug: Flumazenil — Flumazenil- 0.4 mg per 100 µl in a sublingual spray administration
  Other Names: Romzicon,; Anexate®,; BRN 4763661,; Flumazenilo (Spanish),; Flumazenilum (Latin),; Flumazepil; Lanexat®,; Mazicon®,; Ro 151788,; Ro-15-1788,; Romazicon®,; UNII-40P7XK9392
Drug: Placebo — Placebo - only excipients with no API

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of treatment with sublingual (s/l) Flumazenil in healthy volunteers as reversing the effect of the sleep/hypnotic drugs. This study is designed to collect short-term safety and tolerability data.

In addition, the psychomotor/ cognitive and behavioral effects of Flumazenil will be assessed to monitor the degree and the duration of action in a single use of Flumazenil.

ELIGIBILITY:
Inclusion Criteria:

1. The subject understood and voluntarily signed an informed consent form prior to any study-mandated procedure.
2. Male or female aged 18-65 at screening. Women of childbearing potential must have a negative pregnancy test at the screening visit and use a reliable method of contraception during the entire study duration (e.g.

   Contraceptive pill; Intra-uterine device; Contraceptive injection (prolonged-release gestagen); Subdermal implantation;Vaginal ring or Transdermal patch).
3. Body mass index ≥ 18.5 and < 32 kg/m2.
4. Normal sleep habits, i.e. usual self-reported total sleep time > 6 h; usual self-reported time to fall asleep < 30 min; usual bedtime between 10:30 pm and 01:00 am.
5. Subject is in good health as determined by a medical history, physical examination and ECG.
6. Negative any use of illicit drug, alcohol (ethanol), stimulants.

Exclusion Criteria:

1. Any use of medications within 1 month prior to screening visit, except for contraceptive pills.
2. Any sleep associated complains.
3. Previous exposure to Benzodiazepines and/or non-Benzodiazepine hypnotic drugs within 3 months prior to study initiation.
4. History of Epilepsy and or anti-epileptic drugs.
5. Excessive caffeine consumption (≥ 500 mg per day).
6. Pregnancy or breast feeding.
7. Night shift workers within 1 month prior to the screening visit.
8. Clinically relevant ECG abnormalities.
9. History of alcohol or drug abuse within 3 years prior to the screening visit.
10. Cognitive Behavioral Therapy (CBT) started within 1 month prior to the screening visit.
11. Known hypersensitivity to drugs of the same class as the study treatment, or any excipients of the drug formulation.
12. Treatment with another investigational drug within 1 month prior to the screening visit.
13. History of severe head injury.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2010-05; Primary Completion 2012-08 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Safety of single dose administration of sublingual Flumazenil 0.4 mg as a reversal drug for the hypnotic effect of sleep/ hypnotic drugs | 6 months

SECONDARY OUTCOMES:
Efficacy of single dose administration of sublingual Flumazenil 0.4 mg as a reversal drug for the hypnotic effect of sleep/ hypnotic drugs | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Rambam Medical Center, Haifa, Israel